CLINICAL TRIAL: NCT07230691
Title: Prospective, Multi Country, Observational Study of Clinical Outcomes in EGFR-mutated, Advanced Non-Small Cell Lung Cancer (NSCLC) Patients Treated With Approved Amivantamab-containing Regimens Under Standard Clinical Practice
Brief Title: A Study of Clinical Outcomes in Participants With EGFR Mutated Advanced Non-Small Cell Lung Cancer (NSCLC) in a Real-World Setting
Acronym: LEPIDOPTERA
Status: Recruiting | Type: Observational
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 61186372NSC4014; 61186372NSC4014 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2025-11-14; First posted 2025-11-17 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort B: Amivantamab with carboplatin and pemetrexed: Participants with confirmed diagnosis of advanced NSCLC with EGFR exon 19 deletions or exon 21 L858R substitution mutations after failure of prior therapy including an EGFR TKI, who received at least 1 dose of amivantamab in combination with carboplatin and pemetrexed, as per standard clinical practice will be enrolled. No drug will be provided as part of this study. Only data available within routine clinical practice will be collected in this study.
- Cohort C: Amivantamab and lazertinib: Participants with confirmed diagnosis of advanced NSCLC with EGFR exon 19 deletions or exon 21 L858R substitution mutations (first-line therapy) who received at least 1 dose of amivantamab in combination with lazertinib as per standard clinical practice will be enrolled. No drug will be provided as part of this study. Only data available within routine clinical practice will be collected in this study.

SUMMARY:
The purpose of this study is to describe the clinical and health-related outcomes of amivantamab-containing regimens for the treatment of common epidermal growth factor receptor (EGFR) mutated non-small cell lung cancer (NSCLC; most common type of lung cancer) in a real-world setting. Metastatic NSCLC is when this disease spreads to other parts of body. NSCLC may occur due to mutations (changes) in many genes including epidermal growth factor receptor (EGFR).

ELIGIBILITY:
Inclusion Criteria:

* Participant has a confirmed diagnosis of common epidermal growth factor receptor (EGFR)-mutated non-small cell lung cancer (NSCLC) (EGFR exon 19 deletions or exon 21 L858R substitution) and is eligible for an amivantamab-containing regimen per the judgment of the treating physician and in alignment with the approved amivantamab indications and recommended prophylactic and reactive medication as described in the local specific summary of product characteristics (SmPC) for amivantamab
* Participants or their legally acceptable representative, where applicable, must sign a participation agreement/Informed consent form (ICF) allowing source data verification in accordance with local requirements
* Participant is being planned to be initiated with an amivantamab-containing regimen for the first time within 4 weeks following the visit for start of data collection
* Decision to administer an amivantamab-containing regimen has been made prior to participant's enrollment in the study and is separate from the physician's decision to include the participant in the current study

Exclusion criteria:

* At the time of the initiation of the amivantamab-containing regimen, the participant is receiving an active systemic anticancer treatment for advanced NSCLC that is not included in the locally approved combination regimen with amivantamab (regardless of whether it is part of an interventional study). One cycle of platinum-based chemotherapy (for example, carboplatin-pemetrexed) is permitted prior to the first dose of amivantamab in a 1L while awaiting biopsy results
* Participant has received prior treatment with amivantamab in a clinical trial or for compassionate use
* Participants who are not receiving amivantamab but are being treated with a biosimilar or a non-original biologic agent
* Participants with conditions listed in the contraindications of the SmPC for amivantamab or other agents essential for the applicable amivantamab-containing treatment regimen (lazertinib/ platinum/ pemetrexed)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include participants with advanced NSCLC.
Sampling Method: Non-Probability Sample
Enrollment: 380 (Estimated)
Dates: Start 2025-12-03 (Actual); Primary Completion 2030-11-19 (Estimated); Study Completion 2030-12-17 (Estimated)

PRIMARY OUTCOMES:
Real-World Time to Treatment Discontinuation (rwTTD) | Up to approximately 60 Months
  rwTTD is defined as the time from the date of initiation of the amivantamab-containing regimen to discontinuation of the full amivantamab containing regimen for any reason, including disease progression, treatment toxicity or death.

SECONDARY OUTCOMES:
Real-World Progression-Free Survival (rwPFS) | Up to approximately 60 Months
  rwPFS is defined as the time from the date of initiation of the amivantamab-containing regimen to the date of investigator-determined disease progression (radiological or clinical) or death due to any cause, whichever occurs first.
Real-World Time to Next Treatment (rwTTNT) | Up to approximately 60 Months
  rwTTNT is defined as the time from initiation of the amivantamab-containing regimen to start of a subsequent systemic treatment following discontinuation of the full amivantamab-containing regimen or death, whichever occurs first.
Real-World Overall Survival (rwOS) | Up to approximately 60 Months
  rwOS is defined as the time from the date of initiation of the amivantamab-containing regimen to the date of death from any cause or reason.
Real-World Time to Subsequent Treatment Discontinuation (rwTTD2) | Up to approximately 60 Months
  rwTTD2 is defined as the time from initiation of the amivantamab-containing regimen to the discontinuation of the first subsequent therapy for any reason, including disease progression, treatment toxicity or death.
Number of Participants with Adverse Events (AEs) by Severity | Up to approximately 60 Months
  An AE is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.
Number of Participants with Dose Modifications and Discontinuations of Amivantamab, Lazertinib and Chemotherapy | Up to approximately 60 Months
  Participants with Dose Modifications and Discontinuations of Amivantamab, Lazertinib and Chemotherapy will be reported.
Number of Participants Using Concomitant Medications | Up to approximately 60 Months
  Participants using concomitant medications including those to manage specific AEs related to the amivantamab-containing regimen, namely infusion related reactions (IRRs), venous thromboembolism (VTEs), and dermatologic AEs including paronychia, will be reported.
Health-Related Quality of Life (HRQoL) Assessed by SKINDEX Scale Score | Up to approximately 60 Months
  The SKINDEX-16 measures how a participant's skin condition impacts their health-related quality of life. There are 16 questions on a 7-point scale, ranging from 0 (never bothered) to 6 (always bothered). The questionnaire is divided into 3 domains: symptoms (items 1 to 4), emotions (items 5 to 11), and functionality (items 12 to 16). An overall score is the average of the 3 domain scores. All domain scores will be linearly transformed to be in the range from 0 to 100. A score of 0 indicates that the skin condition has no impact on QoL, while a score of 100 indicates the worst possible impact.
Quality of Life Assessed by European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Core Questionnaire (EORTC QLQ-C30) Items-30 Scale Score | Up to approximately 60 Months
  The EORTC QLQ-C30 is a self-administered, 30-item questionnaire measuring the HRQoL of participants with cancer. EORTC QLQ-C30 includes 5 functional scales (physical, role, cognitive, emotional, and social), 3 symptom scales (fatigue, pain, and nausea and vomiting), a global health status / quality of life scale, and 6 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). Responses to items 1-28 are rated on a 4-point Likert response scale ranging from 1 "Not at all" to 4 "Very much." Two global health status items are rated on a 7-point numeric rating scale from 1 "Very Poor" to 7 "Excellent." Higher scores indicate greater functioning, better global health status, and more severe symptoms.
Quality of Life Impact on Questions Regarding Reactive and Prophylactic Management of AEs Related to the Amivantamab-Containing Regimen | Up to approximately 60 Months
  Three questions regarding reactive and prophylactic management of AEs related to the amivantamab-containing regimen will be reported. These questions cover the type of prophylactic/reactive concomitant medication recommended by the treating physician, frequency of use, and the degree of impact on daily life due to use of the respective medication.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (24):
- Klinikum Klagenfurt am Worthersee, Klagenfurt, Austria
- Czechia (2):
  - Fakultni nemocnice Brno, Brno
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
- Germany (7):
  - MVZ am Klinikum Aschaffenburg Onkologie, Aschaffenburg
  - Evangelisches Klinikum Bethel, Bielefeld
  - Klinikum Chemnitz gGmbH, Chemnitz
  - Facharztzentrum Eppendorf, Hamburg
  - Onkologie am Raschplatz, Hanover
  - Klinikum Region Hannover Klinikum Siloah, Hanover
  - Klinikum Konstanz, Konstanz
- Israel (3):
  - Rabin Medical Center, Petah Tikva
  - Sheba Medical Center, Ramat Gan
  - Assuta MC, Tel Aviv
- Italy (11):
  - Oncologia Medica - Irccs - Istituto Tumori Giovanni Paolo II, Bari
  - Istituto di Candiolo, IRCCS, Candiolo
  - Azienda Ospedaliera Pugliese Ciaccio Catanzaro, Catanzaro
  - San Raffaele Hospital, Milan
  - European Institute of Oncology, Milan
  - Fondazione G Pascale Istituto Nazionale Tumori IRCCS, Napoli
  - Azienda Ospedaliero Universitaria Maggiore della Carita di Novara, Novara
  - ASL Gallura - Ospedale Giovanni Paolo II, Olbia
  - Azienda Ospedaliero Universitaria Policlinico Paolo Giaccone, Palermo
  - Azienda Ospedaliero Universitaria di Sassari, Sassari
  - Ospedali Riuniti Di Ancona, Torrette-Ancona

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency